CLINICAL TRIAL: NCT03553394
Title: The Effects on Fluid Balance and Renal Function Using a Restrictive Fluid Strategy in the Postoperative Setting in Patients With Low Urinary Output Undergoing Pancreatic Surgery
Brief Title: Effects of Restrictive Fluid Strategy on Postoperative Oliguric Pancreatic Surgery Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped after interim analysis
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/147
Record Dates: First submitted 2018-05-23; First posted 2018-06-12 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Fluid Therapy; Postoperative Period; Postoperative Complications; Pancreas Disease; Fluid Overload
MeSH Terms: conditions — Postoperative Complications; Pancreatic Diseases; Edema | interventions — Ringer's acetate

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receive a fluid bolus immediately when urinary output is decreased for two consecutive hours or to await fluid bolus therapy for two more hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (Active Comparator): Will receive a fluid bolus 5 ml/kg Ringer's Acetate infusion immediately if oliguric/anuric for two consecutive hours (standard of care).
  Interventions: Drug: Ringer's Acetate
- Expectant management group (No Intervention): Await fluid therapy for 2 hours. Will NOT receive a fluid bolus if oliguric/anuric for two consecutive hours and a now assessment will be made after two more hours.

INTERVENTIONS:
Drug: Ringer's Acetate — Will receive a fluid bolus immediately (Ringer's Acetate 5 mls/kg bw) if oliguric/anuric for two consecutive hours
  Other Names: Ringer Acetate
  Arms: Standard of care group

SUMMARY:
Reduced urinary output is a common postoperative issue for patients going through major surgery such as pancreatic surgery. Commonly this is treated by increasing fluid administration to the patients and sometimes also diuretics. However, overloading patients with fluid also have several risks and known complications. Studies have also shown that a short period of decreased urinary output in the postoperative period do not have an increased incidence of acute renal failure. The aim of our study is to investigate the difference in renal function and postoperative complications associated with fluid overload on these patients that are randomized to either receiving a fluid bolus directly when urinary output decreases or to await for a maximum of four hours to see if urinary output increases spontaneously.

DETAILED DESCRIPTION:
Patents after pancreatic surgery will be included in the study. Oliguric patients (urine output <0.5 ml/kg/h) will be randomized to fluid bolus (5ml/kg Ringer's Acetate in 30 minutes) or no intervention. Primary outcome is difference in urine output two hours after the fluid bolus or no intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients going through pancreatic surgery.

Exclusion Criteria:

* If not oliguric (urinary output <0,5 mls/kg/h) during their stay in the postoperative department
* Hemodynamic instability (the need for >0,1 microgram/kg/min of norepinephrine to keep an acceptable mean arterial pressure based on the patients starting mean arterial pressure).
* Patients that do not want to be a part of the study.
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Urinary output | 2 hours
  Difference in urinary output two hours after giving the patient a fluid bolus (Control Group) or awaiting fluid bolus (interventional Group)..

SECONDARY OUTCOMES:
Renal function | 48 hours
  Renal function after 48 hours
Cumulative fluid balance | 48 hours
  Difference in cumulative fluid balance
Postoperative complications | 90 days
  Frequency of postoperative complications in both groups
Renal replacement therapy | Up to 90 days
  The need for renal replacement therapy during the hospital stay
Mortality | 90 days
  90-day mortality in both groups
Inotropy | 1 week
  Postoperative need of inotropic therapy during the stay in the postoperative department
Vasopressin (ADH) | 1 day
  Levels of vasopressin in serum immediately before and after the operation
S-osmolality | 1 day
  S-osmolality immediately before and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Central ICU (CIVA), Uppsal university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided